## Effects of Awe on Health 11/22/2016

IRB approval date: 11/22/2016

8.25 STATISTICAL METHODS: Briefly summarize the methods and types of analyses that will be performed:

We will conduct multiple regression analyses to determine whether the laboratory measures of emotional reactivity (i.e., ANS reactivity, facial expression, and self-reported experience) are associated with mental health symptoms such as anxiety and depression. We expect that greater negative emotional reactivity as

measured in the laboratory will be associated with worse mood and higher anxiety.

We will use mixed effects models to test whether the awe walk condition had beneficial effects on daily self-reported experience, life satisfaction, and prosociality. We will use analyses of covariance (controlling for age, sex, and education) to examine whether the awe walk condition resulted in decreases in anxiety and depression at the termination of the 8-week intervention and at 3- and 6-months post-intervention.